CLINICAL TRIAL: NCT03073200
Title: Multicenter, Double-Blind, Randomized, Placebo-Controlled Study to Evaluate Safety, Tolerability, and Efficacy of Ixekizumab in Patients From 6 to Less Than 18 Years of Age With Moderate-to-Severe Plaque Psoriasis
Brief Title: Study of Ixekizumab (LY2439821) in Children 6 to Less Than 18 Years With Moderate-to-Severe Plaque Psoriasis
Acronym: Ixora-peds
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 16367; I1F-MC-RHCD (Other: Eli Lilly and Company); 2016-003331-38 (EudraCT Number)
Record Dates: First submitted 2017-03-03; First posted 2017-03-08 (Actual); Results first posted 2020-03-17 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-08-16

CONDITIONS: Plaque Psoriasis
Keywords: children; psoriasis treatment; adolescents
MeSH Terms: interventions — ixekizumab; Etanercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Ixekizumab (Experimental): Ixekizumab given subcutaneously (SC) during the double-blind treatment period and the open-label maintenance period.
  Interventions: Drug: Ixekizumab
- Placebo (Placebo Comparator): Placebo given SC during the double-blind treatment period and then ixekizumab given SC during the open-label maintenance period.
  Interventions: Drug: Placebo
- Open-Label Etanercept (Experimental): Etanercept given SC during the double-blind treatment period and then ixekizumab given SC during the open-label maintenance period. Participants will only be randomized to etanercept in countries where it is approved for severe pediatric psoriasis treatment.
  Interventions: Drug: Etanercept

INTERVENTIONS:
Drug: Ixekizumab — Administered SC
  Other Names: LY2439821
  Arms: Ixekizumab
Drug: Placebo — Administered SC
  Arms: Placebo
Drug: Etanercept — Administered SC
  Arms: Open-Label Etanercept

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of ixekizumab in pediatric participants with moderate-to-severe plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of moderate-to-severe plaque-type psoriasis for at least 6 months prior to baseline as determined by the investigator.
* Have Psoriasis Area and Severity Index (PASI) score ≥12 and a Static Physician Global Assessment (sPGA) ≥3 and body surface area involvement ≥10% at screening and baseline.
* Are candidates for phototherapy or systemic treatment or considered by the investigator as not adequately controlled by topical therapies.
* Male subjects agree to use a reliable method of birth control during the study.
* Female subjects: Participants of childbearing age or childbearing potential who are sexually active who test negative for pregnancy must be counselled and agree to use either 1 highly effective method of contraception or 2 acceptable methods of contraception combined for the duration of the study and for at least 12 weeks following the last dose of study drug, or remain abstinent during the study and for at least 12 weeks following the last dose of study drug.
* Both the child or adolescent and a parent or legal guardian are able to understand and fully participate in the activities of the clinical study and sign their assent and consent, respectively.
* All immunizations are up-to-date in agreement with current immunization guidelines as noted by country specific paediatric authorities (e.g., the American Academy of Paediatrics). Note, subjects who are not up to date or have never been immunized are not to be enrolled in the trial.

Exclusion Criteria:

* Have pustular, erythrodermic, and/or guttate forms of psoriasis.
* Have drug-induced psoriasis.
* Have clinical and/or laboratory evidence of untreated latent or active tuberculosis (TB).
* Participants with a documented history of immune deficiency syndrome.
* Have any other active or recent infection, including chronic or localized infections, within 4 weeks of baseline.
* Subjects with a known history of malignancy, lymphoproliferative disease, including lymphoma, or signs and symptoms suggestive of possible lymphoproliferative disease, such as lymphadenopathy and/or splenomegaly unless ruled out by biopsy.
* Have used any therapeutic agent targeted at reducing interleukin-17.
* Have received other therapies within the specified time frames prior to screening (see below):

  * adalimumab and infliximab 60 days, abatacept 90 days, anakinra 7 days, or any other biologic disease-modifying antirheumatic drug 5 half-lives.
  * systemic therapy for psoriasis and psoriatic arthritis (PsA) (other than above, eg, methotrexate, cyclosporine), phototherapy (eg, photochemotherapy [psoralen plus ultraviolet A]) in the previous 4 weeks.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 201 (Actual)
Dates: Start 2017-03-28 (Actual); Primary Completion 2019-02-07 (Actual); Study Completion 2021-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (69):
- United States (25):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Tien Q. Nguyen, MD inc. DBA First OC Dermatology, Fountain Valley, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Olympian Clinical Research, Clearwater, Florida
  - Solutions Through Advanced Research, Inc., Jacksonville, Florida
  - University of South Florida, Tampa, Florida
  - Forward Clinical Trials, Inc, Tampa, Florida
  - Advanced Medical Research, Sandy Springs, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Arlington Dermatology, Rolling Meadows, Illinois
  - The South Bend Clinic, South Bend, Indiana
  - University of Missouri, Columbia, Missouri
  - SSM Health Cardinal Glennon Children's Hospital, St Louis, Missouri
  - Psoriasis Treatment Center of Central New Jersey, East Windsor, New Jersey
  - University of North Carolina Dermatology and skin Cancer Cen, Chapel Hill, North Carolina
  - Wright State Physicians Dermatology, Fairborn, Ohio
  - Ohio State Univ College Of Medicine, Gahanna, Ohio
  - Oregon Dermatology and Research Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Dermatology and Skin Surgery Center, Exton, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Modern Research Associates PLLC, Dallas, Texas
  - Texas Dermatology and Laser Specialists, San Antonio, Texas
  - Virginia Clinical Research, Norfolk, Virginia
- Argentina (4):
  - Centro de Investigaciones Metabólicas (CINME), Ciudad Autonoma de Buenos Aire, Buenos Aires
  - Fundación Estudios Clínicos- Servicio de Dermatología, Rosario, Santa Fe Province
  - Instituto de Neumonología y Dermatología, Buenos Aires
  - Psoriahue Medicina Interdisciplinaria, Buenos Aires
- Canada (4):
  - Institute for Skin Advancement, Calgary, Alberta
  - Lynderm Research Inc, Markham, Ontario
  - K. Papp Clinical Research Inc, Waterloo, Ontario
  - Hospital Ste Justine, Montreal, Quebec
- Czechia (6):
  - Detska fakultni nemocnice, Brno
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Fakultni Nemocnice Plzen, Plzen-Bory
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - LF UK - Fakultni poliklinika, Prague
  - Nemocnice Na Bulovce, Prague
- France (3):
  - Centre hospitalier universitaire Pellegrin, Bordeaux
  - Hôpital Femme Mère Enfant, Bron
  - CHU de Nice Hopital de L'Archet, Nice
- Germany (5):
  - Universitätsklinikum Erlangen, Erlangen, Bavaria
  - Klinikum der Johann Wolfgang Goethe-Universität Frankfurt, Frankfurt am Main, Hesse
  - Universitätsklinikum Münster, Münster, North Rhine-Westphalia
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz, Rhineland-Palatinate
  - ISA GmbH, Berlin
- Hungary (5):
  - SZTE AOK Borgyogyaszati es Allergologiai Klinika, Szeged, Csongrád megye
  - Debreceni Egyetem Klinikai Kozpont Borgyogyaszati Klinika, Debrecen, Hajdú-Bihar
  - Allergo-Derm Bakos Kft, Szolnok, Jász-Nagykun-Szolnok
  - Szent Janos Korhaz es Eszak-budai Egyesitett Korhazak, Budapest
  - Oroshaza Varosi Onkormanyzat Korhaza, Orosháza
- Mexico (4):
  - Hospital Infantil de Mexico, Mexico City, Federal District
  - Hospital Univ. Dr. Jose Eleuterio Gonzalez, Monterrey, Nuevo León
  - RM Pharma Specialists S.A. de C.V., Distrito Federal
  - Arke Estudios Clinicos S.A. de C.V., Veracruz
- Universitair Medisch Centrum St Radboud Nijmegen, Nijmegen, Netherlands
- Poland (3):
  - "Dermed" Centrum Medyczne Sp. z o.o., Lodz
  - Centralny Szpital Kliniczny MSW, Warsaw
  - DermMEDICA Sp. z o.o., Wroclaw
- Puerto Rico (4):
  - Office of Dr. Samuel Sanchez PSC, Caguas, PR
  - Grupo Dermatologico de Carolina, Carolina, PR
  - Ponce School of Medicine CAIMED Center, Ponce, PR
  - GCM Medical Group PSC, San Juan
- Russia (2):
  - GBUZ Clinical dermatology and venereological dispensary, Krasnodar
  - Center of Children's Health, Moscow
- Spain (3):
  - Hospital Sant Joan de Déu, Esplugues de Llobregat, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Paller AS, Seyger MMB, Magarinos GA, Pinter A, Cather JC, Rodriguez-Capriles C, Zhu D, Somani N, Garrelts A, Papp KA; IXORA-PEDS Investigators. Long-term Efficacy and Safety of Up to 108 Weeks of Ixekizumab in Pediatric Patients With Moderate to Severe Plaque Psoriasis: The IXORA-PEDS Randomized Clinical Trial. JAMA Dermatol. 2022 May 1;158(5):533-541. doi: 10.1001/jamadermatol.2022.0655. PMID 35416908
- See also: Study of Ixekizumab (LY2439821) in Children 6 to Less Than 18 Years With Moderate-to-Severe Plaque Psoriasis — https://trials.lillytrialguide.com/en-US/trial/2xPbhh7bJKOwooYG2OKg6c

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Double-Blind Treatment Period (Week 0 to Week 12), Open-Label Maintenance Period (Week 12 to Week 60), Extension Period (Week 60 to Week 108) followed by post-treatment follow-up period occurring from last treatment visit (week 108), or Early Termination Visit (ETV) for up to 24 weeks following that visit.
  Etanercept (ETN) is reference control group occurred only in Etanercept approved countries.
Pre-assignment Details: The 48-Week Double-Blind, Randomized Withdrawal Period occurs from Week 60 to Week 108 for participants in the Europe who meet the response criterion at Week 60 (defined as sPGA [0,1]).
Groups:
- PBO (Double-Blinded Treatment Period): Participants received matching placebo (PBO) for Ixekizumab (IXE) by subcutaneous injection.
- IXEQ4W (Double-Blinded Treatment Period): Participants with >50 kilogram (kg) weight received 160 milligrams (mg) Ixekizumab at week 0 followed by 80mg Ixekizumab every four weeks (Q4W) from week 4 to 8 followed by 80mg ixekizumab and placebo injection at week 12 by subcutaneous injection.
  Participants with 25 to 50kg received 80mg Ixekizumab at week 0 followed by 40mg Ixekizumab Q4W from week 4 to 8 followed by 40mg ixekizumab and placebo injection at week 12 by subcutaneous injection.
  Participants with >25kg received 40mg Ixekizumab at week 0 followed by 20mg Ixekizumab Q4W from week 4 to 8 followed by 20mg ixekizumab and placebo injection at week 12 by subcutaneous injection.
- ETN (Double-Blinded Treatment Period): Participants received 0.8 milligrams per kilogram (mg/kg) Etanercept (ETN) not exceeding 50mg per dose every week from week 0 to week 11 by subcutaneous injection.
- PBO/IXEQ4W (Maintenance Period); IXEQ4W/IXEQ4W (Maintenance Period); ETN/IXEQ4W (Maintenance Period); PBO/IXEQ4W/IXEQ4W (Extension Period); IXEQ4W/IXEQ4W/IXEQ4W (Extension Period); ETN/IXEQ4W/IXEQ4W (Extension Period): Participants with >50kg received 80mg Ixekizumab every four weeks (Q4W) from week 16 to 56 by subcutaneous injection.
  Participants with 25 to 50kg received 40mg Ixekizumab every four weeks (Q4W) from week 16 to 56 by subcutaneous injection.
  Participants with >25kg received 20mg Ixekizumab every four weeks (Q4W) from week 16 to 56 by subcutaneous injection.
- PBO (Randomized Withdrawal Period): Participants from European Union (EU) countries who meet the response criterion (defined as static Physician's Global Assessment [sPGA] [0,1]) at Week 60 were re-randomized to receive placebo during a 48-Week Double-Blind, Randomized Withdrawal Period.
- IXEQ4W (Randomized Withdrawal Period): Participants from European Union (EU) countries who meet the response criterion (defined as static Physician's Global Assessment [sPGA] [0,1]) at Week 60 were re-randomized to ixekizumab 20, 40, or 80 mg every 4 weeks (Q4W) according to their weight at the time of rerandomization during a 48-Week Double-Blind, Randomized Withdrawal Period.
- IXEQ4W_Re-Treatment (Randomized Withdrawal) Period: Participants from EU countries who do not meet the response criterion at Week 60 continued with open-label treatment with ixekizumab.
- PBO (Post-Treatment Follow-Up); IXEQ4W (Post-Treatment Follow-Up); ETN (Post-Treatment Follow-Up): Participants who received study drug including those who discontinue the study, were monitored at approximately 4 and 12 weeks after the date of their final injection of study drug to monitor clinical safety, including neutrophil levels.
Period: Double Blind Treatment Period
Arm/Group | PBO (Double-Blinded Treatment Period) | IXEQ4W (Double-Blinded Treatment Period) | ETN (Double-Blinded Treatment Period) | PBO/IXEQ4W (Maintenance Period) | IXEQ4W/IXEQ4W (Maintenance Period) | ETN/IXEQ4W (Maintenance Period) | PBO/IXEQ4W/IXEQ4W (Extension Period) | IXEQ4W/IXEQ4W/IXEQ4W (Extension Period) | ETN/IXEQ4W/IXEQ4W (Extension Period) | PBO (Randomized Withdrawal Period) | IXEQ4W (Randomized Withdrawal Period) | IXEQ4W_Re-Treatment (Randomized Withdrawal) Period | PBO (Post-Treatment Follow-Up) | IXEQ4W (Post-Treatment Follow-Up) | ETN (Post-Treatment Follow-Up)
Started | 56 | 115 | 30 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Participants in Etanercept Approved Countries | 19 | 38 | 30 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 54 | 114 | 30 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Parent/Guardian | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Open-Label Maintenance Period
Arm/Group | PBO (Double-Blinded Treatment Period) | IXEQ4W (Double-Blinded Treatment Period) | ETN (Double-Blinded Treatment Period) | PBO/IXEQ4W (Maintenance Period) | IXEQ4W/IXEQ4W (Maintenance Period) | ETN/IXEQ4W (Maintenance Period) | PBO/IXEQ4W/IXEQ4W (Extension Period) | IXEQ4W/IXEQ4W/IXEQ4W (Extension Period) | ETN/IXEQ4W/IXEQ4W (Extension Period) | PBO (Randomized Withdrawal Period) | IXEQ4W (Randomized Withdrawal Period) | IXEQ4W_Re-Treatment (Randomized Withdrawal) Period | PBO (Post-Treatment Follow-Up) | IXEQ4W (Post-Treatment Follow-Up) | ETN (Post-Treatment Follow-Up)
Started | 0 (This period is to report Maintenance Period participants.) | 0 (This period is to report Maintenance Period participants.) | 0 (This period is to report Maintenance Period participants.) | 53 (This period is to report Maintenance Period participants.) | 113 (This period is to report Maintenance Period participants.) | 28 (This period is to report Maintenance Period participants.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 49 | 109 | 28 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 4 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Participant moved to another city | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Extension Period
Arm/Group | PBO (Double-Blinded Treatment Period) | IXEQ4W (Double-Blinded Treatment Period) | ETN (Double-Blinded Treatment Period) | PBO/IXEQ4W (Maintenance Period) | IXEQ4W/IXEQ4W (Maintenance Period) | ETN/IXEQ4W (Maintenance Period) | PBO/IXEQ4W/IXEQ4W (Extension Period) | IXEQ4W/IXEQ4W/IXEQ4W (Extension Period) | ETN/IXEQ4W/IXEQ4W (Extension Period) | PBO (Randomized Withdrawal Period) | IXEQ4W (Randomized Withdrawal Period) | IXEQ4W_Re-Treatment (Randomized Withdrawal) Period | PBO (Post-Treatment Follow-Up) | IXEQ4W (Post-Treatment Follow-Up) | ETN (Post-Treatment Follow-Up)
Started | 0 | 0 | 0 | 0 (This period is to report Extension Period participants.) | 0 (This period is to report Extension Period participants.) | 0 (This period is to report Extension Period participants.) | 34 (This period is to report Extension Period participants.) | 68 (This period is to report Extension Period participants.) | 9 (This period is to report Extension Period participants.) | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 31 | 62 | 7 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 6 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Sponsor Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Parent/Guardian | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Randomized Withdrawal Period
Arm/Group | PBO (Double-Blinded Treatment Period) | IXEQ4W (Double-Blinded Treatment Period) | ETN (Double-Blinded Treatment Period) | PBO/IXEQ4W (Maintenance Period) | IXEQ4W/IXEQ4W (Maintenance Period) | ETN/IXEQ4W (Maintenance Period) | PBO/IXEQ4W/IXEQ4W (Extension Period) | IXEQ4W/IXEQ4W/IXEQ4W (Extension Period) | ETN/IXEQ4W/IXEQ4W (Extension Period) | PBO (Randomized Withdrawal Period) | IXEQ4W (Randomized Withdrawal Period) | IXEQ4W_Re-Treatment (Randomized Withdrawal) Period | PBO (Post-Treatment Follow-Up) | IXEQ4W (Post-Treatment Follow-Up) | ETN (Post-Treatment Follow-Up)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 (This period is to report randomized withdrawal period participants.) | 0 (This period is to report randomized withdrawal period participants.) | 0 (This period is to report randomized withdrawal period participants.) | 33 (This period is to report randomized withdrawal period participants.) | 34 (This period is to report randomized withdrawal period participants.) | 33 (This period is to report randomized withdrawal period participants.) | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 33 | 32 | 30 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Parent/Guardian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Period: Post-Treatment Follow-Up Period
Arm/Group | PBO (Double-Blinded Treatment Period) | IXEQ4W (Double-Blinded Treatment Period) | ETN (Double-Blinded Treatment Period) | PBO/IXEQ4W (Maintenance Period) | IXEQ4W/IXEQ4W (Maintenance Period) | ETN/IXEQ4W (Maintenance Period) | PBO/IXEQ4W/IXEQ4W (Extension Period) | IXEQ4W/IXEQ4W/IXEQ4W (Extension Period) | ETN/IXEQ4W/IXEQ4W (Extension Period) | PBO (Randomized Withdrawal Period) | IXEQ4W (Randomized Withdrawal Period) | IXEQ4W_Re-Treatment (Randomized Withdrawal) Period | PBO (Post-Treatment Follow-Up) | IXEQ4W (Post-Treatment Follow-Up) | ETN (Post-Treatment Follow-Up)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 (This period is to report Follow-Up period participants.) | 0 (This period is to report Follow-Up period participants.) | 0 (This period is to report Follow-Up period participants.) | 6 (This period is to report Follow-Up period participants.) | 166 (This period is to report Follow-Up period participants.) | 2 (This period is to report Follow-Up period participants.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 139 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 27 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Participant moved to another city | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Site terminated by sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Parent/Guardian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 0
Not completed — Other-determined by Investigator | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Participants received matching placebo for Ixekizumab by subcutaneous injection.
- Ixekizumab: Participants with >50kg received 160mg Ixekizumab at week 0 followed by 80mg Ixekizumab Q4W from week 4 to 8 followed by 80mg ixekizumab and placebo injection at week 12 by subcutaneous injection.
  Participants with 25 to 50kg received 80mg Ixekizumab at week 0 followed by 40mg Ixekizumab Q4W from week 4 to 8 followed by 40mg ixekizumab and placebo injection at week 12 by subcutaneous injection.
  Participants with >25kg received 40mg Ixekizumab at week 0 followed by 20mg Ixekizumab Q4W from week 4 to 8 followed by 20mg ixekizumab and placebo injection at week 12 by subcutaneous injection.
- Open-label Etanercept: Participants received 0.8mg/kg Etanercept not exceeding 50mg per dose every week from week 0 to week 11 by subcutaneous injection.
- Total: Total of all reporting groups
Arm/Group | Placebo | Ixekizumab | Open-label Etanercept | Total
Number analyzed (Participants) | 56 | 115 | 30 | 201
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.1 (2.79) | 13.7 (3.14) | 13.7 (2.95) | 13.5 (3.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 63 | 18 | 117
  Male | 20 | 52 | 12 | 84
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 30 | 7 | 48
  Not Hispanic or Latino | 42 | 82 | 23 | 147
  Unknown or Not Reported | 3 | 3 | 0 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 1 | 3
  Asian | 2 | 4 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 3 | 0 | 6
  White | 45 | 95 | 25 | 165
  More than one race | 3 | 10 | 3 | 16
  Unknown or Not Reported | 3 | 1 | 1 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  Puerto Rico | 3 | 5 | 0 | 8
  Argentina | 3 | 7 | 3 | 13
  Hungary | 6 | 13 | 2 | 21
  United States | 22 | 42 | 0 | 64
  Czechia | 2 | 6 | 4 | 12
  Spain | 5 | 4 | 3 | 12
  Russia | 4 | 7 | 4 | 15
  Canada | 1 | 6 | 0 | 7
  Netherlands | 0 | 1 | 0 | 1
  Poland | 5 | 12 | 8 | 25
  Mexico | 1 | 4 | 2 | 7
  France | 1 | 1 | 1 | 3
  Germany | 3 | 7 | 3 | 13
Psoriasis Area Severity Index (PASI) [Mean (Standard Deviation); unit: Score on a scale] — PASI combines assessments of the extent of body surface involvement in 4 regions (head & neck(h), trunk(t), arms(u), legs(l)) & severity of scaling (S), redness (R), & plaque induration/infiltration (thickness, T) in each region. Severity is rated for each index (R, S, T) on a 0-4 scale (0 for no involvement up to 4 for severe involvement): 0 = none, 1 = slight, 2 = mild, 3 = moderate, 4 = severe Fraction of total body surface area affected is graded on a 0-6 scale (0 for no involvement to 6 for 90% - 100% involvement).
  Overall score ranges from 0 (no psoriasis) to 72 (most severe disease).
  Score on a scale | 19.73 (8.010) | 19.75 (7.509) | 24.78 (7.448) | 20.49 (7.81)
(sPGA) [Mean (Standard Deviation); unit: Score on a scale] — Static Physician Global Assessment (sPGA): The physician's global assessment of the Participant's psoriasis lesions at a given time point. Plaques are assessed for induration, erythema, and scaling, and an overall rating of psoriasis severity is given using the anchors of clear (0), minimal (1), mild (2), moderate (3), severe (4), or very severe (5).
  Score on a scale | 3.5 (0.63) | 3.6 (0.61) | 4.1 (0.31) | 3.63 (0.61)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a ≥75% Improvement in Psoriasis Area and Severity Index (PASI 75) (Placebo and Ixekizumab)
Description: PASI combines assessments of the extent of body surface involvement in 4 regions (head & neck(h), trunk(t), arms(u), legs(l)) & severity of scaling (S), redness (R), & plaque induration/infiltration (thickness, T) in each region. Severity is rated for each index (R, S, T) on a 0-4 scale (0 for no involvement up to 4 for severe involvement): 0 = none, 1 = slight, 2 = mild, 3 = moderate, 4 = severe Fraction of total body surface area (BSA) affected is graded on a 0-6 scale (0 for no involvement to 6 for 90% - 100% involvement): 0 = 0% (clear), 1 = >0% to <10%, 2 = 10% to <30%, 3 = 30% to <50%, 4 = 50% to <70%, 5 = 70% to 90%, 6 = 90% to 100%.
  Overall score ranges from 0 (no psoriasis) to 72 (most severe disease).
Time Frame: Week 12
Population: All randomized Participants in placebo and Ixekizumab arms. Missing values were imputed by Nonresponder imputation.
  Participants who do not meet the clinical response criteria or have missing clinical response data or without at least 1 post-baseline observation are considered as nonresponders for NRI analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ixekizumab
Number analyzed (Participants) | 56 | 115
percentage of participants | 25 | 88.7
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab; Test type: Superiority; p < 0.001, Fisher Exact; Mean Difference (Final Values) = 63.7, 95% CI 2-sided [51.0 to 76.4]

2. Primary Outcome: Percentage of Participants With a Static Physician Global Assessment (sPGA) (0,1) (Placebo and Ixekizumab)
Description: Static Physician Global Assessment (sPGA): The physician's global assessment of the Participant's psoriasis lesions at a given time point. Plaques are assessed for induration, erythema, and scaling, and an overall rating of psoriasis severity is given using the anchors of clear (0), minimal (1), mild (2), moderate (3), severe (4), or very severe (5). An sPGA assessed as either 0 or 1 represents a clinically meaningful response of minimal plaque severity or complete resolution of plaque psoriasis.
Time Frame: Week 12
Population: All randomized participants in placebo and Ixekizumab arms. Missing values were imputed by Nonresponder imputation(NRI).
  Pts who do not meet the clinical response criteria or have missing clinical response data or without at least 1 post-baseline observation are considered as nonresponders for NRI analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ixekizumab
Number analyzed (Participants) | 56 | 115
percentage of participants | 10.7 | 80.9
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab; Test type: Superiority; p < 0.001, Fisher Exact; Mean Difference (Final Values) = 70.2, 95% CI 2-sided [59.3 to 81]

3. Secondary Outcome: Percentage of Participants With a ≥90% Improvement in Psoriasis Area and Severity Index (PASI 90)
Description: PASI combines assessments of the extent of body surface involvement in 4 regions (head & neck(h), trunk(t), arms(u), legs(l)) & severity of scaling (S), redness (R), & plaque induration/infiltration (thickness, T) in each region. Severity is rated for each index (R, S, T) on a 0-4 scale (0 for no involvement up to 4 for severe involvement): 0 = none, 1 = slight, 2 = mild, 3 = moderate, 4 = severe Fraction of total BSA affected is graded on a 0-6 scale (0 for no involvement to 6 for 90% - 100% involvement): 0 = 0% (clear), 1 = >0% to <10%, 2 = 10% to <30%, 3 = 30% to <50%, 4 = 50% to <70%, 5 = 70% to 90%, 6 = 90% to 100%.Overall score ranges from 0 (no psoriasis) to 72 (most severe disease).
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ixekizumab
Number analyzed (Participants) | 56 | 115
percentage of participants | 5.4 | 78.3
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab; Test type: Superiority; p < 0.001, Fisher Exact; Mean Difference (Final Values) = 72.9, 95% CI 2-sided [63.3 to 82.5]

4. Secondary Outcome: Percentage of Participants With a sPGA (0)
Description: Static Physician Global Assessment (sPGA): The physician's global assessment of the Participant's psoriasis lesions at a given time point. Plaques are assessed for induration, erythema, and scaling, and an overall rating of psoriasis severity is given using the anchors of clear (0), minimal (1), mild (2), moderate (3), severe (4), or very severe (5). An sPGA assessed as either 0 or 1 represents a clinically meaningful response of minimal plaque severity or complete resolution of plaque psoriasis.
  An sPGA assessed as 0 represents a clinically important endpoint indicating complete resolution of plaque psoriasis.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ixekizumab
Number analyzed (Participants) | 56 | 115
percentage of participants | 1.8 | 52.2
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab; Test type: Superiority; p < 0.001, Fisher Exact; Mean Difference (Final Values) = 50.4, 95% CI 2-sided [40.6 to 60.2]

5. Secondary Outcome: Percentage of Participants With a 100% Improvement in Psoriasis Area and Severity Index (PASI 100)
Description: PASI combines assessments of the extent of body surface involvement in 4 regions (head & neck(h), trunk(t), arms(u), legs(l)) & severity of scaling (S), redness (R), & plaque induration/infiltration (thickness, T) in each region. Severity is rated for each index (R, S, T) on a 0-4 scale (0 for no involvement up to 4 for severe involvement): 0 = none, 1 = slight, 2 = mild, 3 = moderate, 4 = severe Fraction of total BSA affected is graded on a 0-6 scale (0 for no involvement to 6 for 90% - 100% involvement): 0 = 0% (clear), 1 = >0% to <10%, 2 = 10% to <30%, 3 = 30% to <50%, 4 = 50% to <70%, 5 = 70% to 90%, 6 = 90% to 100%.
  Overall score ranges from 0 (no psoriasis) to 72 (most severe disease).
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ixekizumab
Number analyzed (Participants) | 56 | 115
percentage of participants | 1.8 | 49.6
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab; Test type: Superiority; p < 0.001, Fisher Exact; Mean Difference (Final Values) = 47.8, 95% CI 2-sided [38.0 to 57.6]

6. Secondary Outcome: Percentage of Participants With a ≥75% Improvement in Psoriasis Area and Severity Index (PASI 75)
Description: as for outcome 5
Time Frame: Week 4
Population: All randomized participants in placebo and Ixekizumab arms. Missing values were imputed by Nonresponder imputation.
  Pts who do not meet the clinical response criteria or have missing clinical response data or without at least 1 post-baseline observation are considered as nonresponders for NRI analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ixekizumab
Number analyzed (Participants) | 56 | 115
percentage of participants | 8.9 | 53.9
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab; Test type: Superiority; p < 0.001, Fisher Exact; Mean Difference (Final Values) = 45, 95% CI 2-sided [33.2 to 56.8]

7. Secondary Outcome: Percentage of Participants With a Static Physician Global Assessment (sPGA) (0,1)
Description: as for outcome 2
Time Frame: Week 4
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ixekizumab
Number analyzed (Participants) | 56 | 115
percentage of participants | 7.1 | 47.8
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab; Test type: Superiority; p < 0.001, Fisher Exact; Mean Difference (Final Values) = 40.7, 95% CI 2-sided [29.3 to 52.0]

8. Secondary Outcome: Percentage of Participants With an Improvement of ≥4 in Those Who Had a Baseline Itch Numeric Rating Scale (NRS) Score of ≥4
Description: Itch Numeric Rating Scale (NRS): is a single-item, patient-reported outcome (PRO) measure designed to capture the overall severity of a participant's itching due to his/her psoriasis by having the patient circle the integer that describes the worst level of itching in the past 24 hours on an 11-point NRS anchored at 0 representing "no itching" and 10 representing "worst itch imaginable.
Time Frame: Week 12
Population: All randomized participants with baseline Itch NRS Score >=4 in placebo and Ixekizumab arms.
  Missing values were imputed by NRI. Participants who do not meet the clinical response criteria or have missing clinical response data or without at least 1 post-baseline observation are considered as nonresponders for NRI analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ixekizumab
Number analyzed (Participants) | 40 | 83
percentage of participants | 20.0 | 71.1
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab; Test type: Superiority; p < 0.001, Fisher Exact; Mean Difference (Final Values) = 51.1, 95% CI 2-sided [35.3 to 66.9]

9. Secondary Outcome: Percentage of Participants Achieving Children's Dermatology Life Quality Index (CDLQI)/Dermatology Life Quality Index (DLQI) (0/1)
Description: DLQI is a validated, dermatology-specific, patient reported measure that evaluates participant's health-related quality of life. It consists of 10 items that are grouped in 6 domains: symptoms & feelings, daily activities, leisure, work & school , personal relationships, & treatment. The recall period of this scale is over the "last week." Response categories and corresponding scores are:
  Very much = 3, A lot = 2, A little = 1, Not at all = 0, Not relevant = 0. A DLQI total score is calculated by summing all 10 items responses, and has a range of 0 to 30 (higher scores are indicative of greater impairment). CDLQI questionnaire is designed for use in children (4 to 16 years of age). It consists of 10 items that are grouped into 6 domains: symptoms & feelings, leisure, school or holidays, personal relationships, sleep, & treatment. A CDLQI total score is calculated by summing all 10 items responses, and has a range of 0 to 30 (higher scores are indicative of greater impairment).
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ixekizumab
Number analyzed (Participants) | 56 | 115
percentage of participants | 23.2 | 64.3
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab; Test type: Superiority; p < 0.001, Fisher Exact; Mean Difference (Final Values) = 41.1, 95% CI 2-sided [27.0 to 55.2]

10. Secondary Outcome: Change From Baseline on the Nail Psoriasis Severity Index (NAPSI)
Description: NAPSI is a numeric, reproducible, objective tool for evaluation of nail psoriasis. This scale was used to evaluate the severity of nail bed psoriasis & nail matrix psoriasis by area of involvement in the nail unit. Both fingernail & toenail involvement were assessed.The nail is divided with imaginary horizontal & longitudinal lines into quadrants. Each nail is given a score for nail bed psoriasis (0 to 4) & nail matrix psoriasis (0 to 4), depending on the presence (score of 1) or absence (score of 0) of any of the features of nail bed & nail matrix psoriasis in each quadrant:
  0 = None
  1. = present in one quadrant of nail
  2. = present in two quadrants of nail
  3. = present in three quadrants of nail
  4. = present in four quadrants of nail NAPSI score of a nail is the sum of scores in nail bed & nail matrix from each quadrant (maximum of 8). Each nail is evaluated, & the sum of all the fingernails and toenails is the total NAPSI score ranging from 0 to 160 (No to Severe nail Psoriasis)
Time Frame: Baseline, Week 12
Population: All randomized participants with baseline and post baseline NAPSI score in placebo and Ixekizumab arms.
  Least squares(LS) Mean was calculated using mixed model repeated measures (MMRM) with treatment, region, baseline sPGA score,baseline weight category, baseline value, visit, treatment-by-visit, & baseline-by-visit interactions as fixed factors.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Ixekizumab
Number analyzed (Participants) | 12 | 34
score on a scale | 0.17 (5.331) | -16.87 (3.110)
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab; Test type: Superiority; p = 0.005, Mixed Models Analysis; Mean Difference (Final Values) = -17.04, 95% CI 2-sided [-28.70 to -5.38], Standard Error of Mean 5.747

11. Secondary Outcome: Change From Baseline on the Psoriasis Scalp Severity Index (PSSI)
Description: The scalp was assessed for erythema (redness), induration (hardness), and desquamation (shedding of skin) and percentage of area affected as follows:
  Erythema, Induration and Desquamation:
  0 = Absent
  1. = Slight
  2. = Moderate
  3. = Severe
  4. = Severest Possible
  Percent of Scalp Involved:
  1. = <10%
  2. = 10% - 29%
  3. = 30% - 49%
  4. = 50% - 69%
  5. = 70% - 89%
  6. = 90% - 100%
  The PSSI score is a composite score derived from the sum of the scores for erythema, induration and desquamation multiplied by the score for the extent of scalp area involved (percent of scalp involved). The range is 0 (no psoriasis) to 72 (Most severe Disease).
  LSMean was calculated using treatment, region, baseline sPGA score, baseline weight category, baseline value, visit, treatment-by-visit, and baseline-by-visit interactions as fixed factors.
Time Frame: Baseline, Week 12
Population: All randomized participants with baseline and post-baseline PSSI score in placebo and Ixekizumab.
  LSMean was calculated using MMRM model with treatment, region, baseline sPGA score, baseline weight category, baseline value, visit, treatment-by-visit, and baseline-by-visit interactions as fixed factors.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Ixekizumab
Number analyzed (Participants) | 50 | 102
score on a scale | -12.28 (2.572) | -27.64 (2.320)
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -15.36, 95% CI 2-sided [-18.69 to -12.04], Standard Error of Mean 1.682

12. Secondary Outcome: Change From Baseline on the Palmoplantar Psoriasis Severity Index (PPASI)
Description: PPASI was used if the participant has palmoplantar psoriasis at baseline. Both the palms & soles on each hand & foot was assessed for erythema, induration, desquamation & percentage of area affected as follows:
  Erythema (E), Induration (I), & Desquamation (D):0 = None, 1 = Slight, 2 = Moderate, 3 = Severe, 4 = Very Severe
  Percent of Palm and Sole Area Covered:
  0 = None, 1 = <10%, 2 = 10% - 29%, 3 = 30% - 49%, 4 = 50% - 69%, 5 = 70% - 89%, 6 = 90% - 100% PPASI score is a composite score derived from the sum scores for E, I, & D multiplied by a score for the extent of palm & sole area involvement. The range is 0 (no psoriasis) to 72 (most severe disease).
Time Frame: Baseline, Week 12
Population: All randomized participants with baseline PPASI score in placebo and Ixekizumab arms.
  LSMean was calculated using MMRM model with treatment, region, baseline sPGA score, baseline weight category, baseline value, visit, treatment-by-visit, and baseline-by-visit interactions as fixed factors.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Ixekizumab
Number analyzed (Participants) | 9 | 17
score on a scale | 6.89 (3.37) | -5.11 (2.148)
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab; Test type: Superiority; p = 0.006, Mixed Models Analysis; Mean Difference (Final Values) = -12.01, 95% CI 2-sided [-20.11 to -3.90], Standard Deviation 3.853

13. Secondary Outcome: Number of Participants With Anti-Ixekizumab Antibodies
Description: A treatment emergent - antidrug antibody (TE-ADA) positive participant were defined as:
  1. a participant with a >= 4-fold increase over a positive baseline antibody titer; or
  2. for a negative baseline titer, a participant with an increase from the baseline to a level of >= 1:10.
Time Frame: Baseline through Week 48
Population: All randomized participants from maintenance period (During maintenance period participants were on Ixekizumab treatment).
Measure: Number; unit: participants
Groups:
- Ixekizumab (Maintenance Period): Participants with >50kg received 80mg Ixekizumab every four weeks (Q4W) from week 16 to 56 by subcutaneous injection.
  Participants with 25 to 50kg received 40mg Ixekizumab every four weeks (Q4W) from week 16 to 56 by subcutaneous injection.
  Participants with >25kg received 20mg Ixekizumab every four weeks (Q4W) from week 16 to 56 by subcutaneous injection.
Arm/Group | Ixekizumab (Maintenance Period)
Number analyzed (Participants) | 194
participants | 56

14. Secondary Outcome: Pharmacokinetics (PK): Trough Ixekizumab Concentration at Steady State (Ctrough ss)
Description: Pharmacokinetics (PK): Trough Ixekizumab Concentration at Steady State (Ctrough ss).
Time Frame: Week 12
Population: All randomized participants in Ixekizumab arm with week 12 PK samples.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (μg/mL)
Arm/Group | Ixekizumab
Number analyzed (Participants) | 111
microgram per milliliter (μg/mL) | 3.03 (106)

15. Secondary Outcome: Percentage of Participants With a ≥75% Improvement in Psoriasis Area and Severity Index (PASI 75) (Etanercept Approved Countries)
Description: as for outcome 5
Time Frame: Week 12
Population: All randomized participants in Etanercept approved countries per protocol addendum. Missing values were imputed by Nonresponder imputation.
  Participants who do not meet the clinical response criteria or have missing clinical response data or without at least 1 post-baseline observation are considered as nonresponders for NRI analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ixekizumab | Open-Label Etanercept
Number analyzed (Participants) | 19 | 38 | 30
percentage of participants | 26.3 | 84.2 | 63.3
Statistical Analysis 1: Comparison: Ixekizumab vs Open-Label Etanercept; Test type: Superiority; p = 0.089, Fisher Exact; Mean Difference (Final Values) = 20.9, 95% CI 2-sided [0.1 to 41.7]

16. Secondary Outcome: Percentage of Participants With a Static Physician Global Assessment (sPGA) (0,1) (Etanercept Approved Countries)
Description: as for outcome 2
Time Frame: Week 12
Population: as for outcome 15
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ixekizumab | Open-Label Etanercept
Number analyzed (Participants) | 19 | 38 | 30
percentage of participants | 5.3 | 76.3 | 53.3
Statistical Analysis 1: Comparison: Ixekizumab vs Open-Label Etanercept; Test type: Superiority; p = 0.070, Fisher Exact; Mean Difference (Final Values) = 23.0, 95% CI 2-sided [0.6 to 45.4]

ADVERSE EVENTS:
Time Frame: Up to 132 Weeks
Description: All randomized participants who received at least one dose of study drug. There are gender specific adverse events, only occurring in male or female participants. The number of participants exposed has been adjusted accordingly.
Groups:
- PBO (Double-Blinded Treatment Period): Participants received matching placebo for Ixekizumab by subcutaneous injection.
- IXEQ4W (Double-Blinded Treatment Period): Participants with >50kg received 160mg Ixekizumab at week 0 followed by 80mg Ixekizumab every four weeks (Q4W) from week 4 to 8 followed by 80mg ixekizumab and placebo injection at week 12 by subcutaneous injection.
  Participants with 25 to 50kg received 80mg Ixekizumab at week 0 followed by 40mg Ixekizumab Q4W from week 4 to 8 followed by 40mg ixekizumab and placebo injection at week 12 by subcutaneous injection.
  Participants with >25kg received 40mg Ixekizumab at week 0 followed by 20mg Ixekizumab Q4W from week 4 to 8 followed by 20mg ixekizumab and placebo injection at week 12 by subcutaneous injection.
- ETN (Double-Blinded Treatment Period): Participants received 0.8mg/kg Etanercept not exceeding 50mg per dose every week from week 0 to week 11 by subcutaneous injection.
- IXEQ4W_Re-Treatment (Randomized Withdrawal) Period: Participants from EU countries who do not meet the response criterion at Week 60 will continue with open-label treatment with ixekizumab.
- PBO (Post-Treatment Follow-Up); IXEQ4W (Post-Treatment Follow-Up); ETN (Post-Treatment Follow-Up): Participants who received study drug including those who discontinue the study, will be monitored at approximately 4 and 12 weeks after the date of their final injection of study drug to monitor clinical safety, including neutrophil levels.
Arm/Group | PBO (Double-Blinded Treatment Period) | IXEQ4W (Double-Blinded Treatment Period) | ETN (Double-Blinded Treatment Period) | PBO/IXEQ4W (Maintenance Period) | IXEQ4W/IXEQ4W (Maintenance Period) | ETN/IXEQ4W (Maintenance Period) | PBO/IXEQ4W/IXEQ4W (Extension Period) | IXEQ4W/IXEQ4W/IXEQ4W (Extension Period) | ETN/IXEQ4W/IXEQ4W (Extension Period) | PBO (Randomized Withdrawal Period) | IXEQ4W (Randomized Withdrawal Period) | IXEQ4W_Re-Treatment (Randomized Withdrawal) Period | PBO (Post-Treatment Follow-Up) | IXEQ4W (Post-Treatment Follow-Up) | ETN (Post-Treatment Follow-Up)
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/115 | 0/30 | 0/53 | 0/113 | 0/28 | 0/34 | 0/68 | 0/9 | 0/33 | 0/34 | 0/33 | 0/6 | 0/166 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/56 | 1/115 | 1/30 | 3/53 | 7/113 | 1/28 | 0/34 | 2/68 | 0/9 | 0/33 | 3/34 | 0/33 | 0/6 | 1/166 | 0/2
Other Adverse Events (participants affected / at risk) | 14/56 | 49/115 | 7/30 | 33/53 | 76/113 | 18/28 | 20/34 | 43/68 | 5/9 | 15/33 | 22/34 | 11/33 | 2/6 | 9/166 | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | PBO (Double-Blinded Treatment Period) (N=56) | IXEQ4W (Double-Blinded Treatment Period) (N=115) | ETN (Double-Blinded Treatment Period) (N=30) | PBO/IXEQ4W (Maintenance Period) (N=53) | IXEQ4W/IXEQ4W (Maintenance Period) (N=113) | ETN/IXEQ4W (Maintenance Period) (N=28) | PBO/IXEQ4W/IXEQ4W (Extension Period) (N=34) | IXEQ4W/IXEQ4W/IXEQ4W (Extension Period) (N=68) | ETN/IXEQ4W/IXEQ4W (Extension Period) (N=9) | PBO (Randomized Withdrawal Period) (N=33) | IXEQ4W (Randomized Withdrawal Period) (N=34) | IXEQ4W_Re-Treatment (Randomized Withdrawal) Period (N=33) | PBO (Post-Treatment Follow-Up) (N=6) | IXEQ4W (Post-Treatment Follow-Up) (N=166) | ETN (Post-Treatment Follow-Up) (N=2)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inflammatory bowel disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster oticus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis media acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative ileus (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Splenic rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glucose tolerance decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0/36 (0) | 0/63 (0) | 0/18 (0) | 1/35 (1) | 0/61 (0) | 0/17 (0) | 0/22 (0) | 0/37 (0) | 0/3 (0) | 0/17 (0) | 0/23 (0) | 0/19 (0) | 0/2 (0) | 0/104 (0) | 0/1 (0)
Renal haematoma (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0/36 (0) | 0/63 (0) | 0/18 (0) | 0/35 (0) | 1/61 (1) | 0/17 (0) | 0/22 (0) | 0/37 (0) | 0/3 (0) | 0/17 (0) | 0/23 (0) | 0/19 (0) | 0/2 (0) | 0/104 (0) | 0/1 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | PBO (Double-Blinded Treatment Period) (N=56) | IXEQ4W (Double-Blinded Treatment Period) (N=115) | ETN (Double-Blinded Treatment Period) (N=30) | PBO/IXEQ4W (Maintenance Period) (N=53) | IXEQ4W/IXEQ4W (Maintenance Period) (N=113) | ETN/IXEQ4W (Maintenance Period) (N=28) | PBO/IXEQ4W/IXEQ4W (Extension Period) (N=34) | IXEQ4W/IXEQ4W/IXEQ4W (Extension Period) (N=68) | ETN/IXEQ4W/IXEQ4W (Extension Period) (N=9) | PBO (Randomized Withdrawal Period) (N=33) | IXEQ4W (Randomized Withdrawal Period) (N=34) | IXEQ4W_Re-Treatment (Randomized Withdrawal) Period (N=33) | PBO (Post-Treatment Follow-Up) (N=6) | IXEQ4W (Post-Treatment Follow-Up) (N=166) | ETN (Post-Treatment Follow-Up) (N=2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 6 (6) | 0 (0) | 1 (1) | 3 (5) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 5 (7) | 0 (0) | 3 (3) | 5 (6) | 1 (1) | 1 (1) | 3 (7) | 0 (0) | 1 (1) | 2 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 6 (6) | 0 (0) | 3 (3) | 8 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 5 (5) | 0 (0) | 3 (3) | 7 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 11 (16) | 0 (0) | 8 (16) | 20 (47) | 0 (0) | 0 (0) | 2 (6) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 4 (6) | 1 (1) | 4 (4) | 4 (5) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 4 (5) | 6 (7) | 1 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Impetigo (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 7 (13) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 4 (5) | 0 (0) | 1 (1) | 4 (5) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 4 (4) | 13 (15) | 0 (0) | 7 (9) | 16 (21) | 4 (6) | 0 (0) | 8 (10) | 0 (0) | 4 (4) | 11 (14) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 2 (3) | 8 (12) | 4 (4) | 3 (3) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 5 (5) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 5 (9) | 4 (5) | 1 (1) | 4 (5) | 0 (0) | 1 (1) | 3 (3) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 6 (7) | 0 (0) | 5 (8) | 13 (20) | 2 (2) | 10 (13) | 11 (13) | 0 (0) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 4 (4) | 3 (4) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 2 (3) | 4 (4) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 6 (6) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 3 (4) | 4 (5) | 3 (3) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 7 (8) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (2) | 12 (13) | 1 (1) | 2 (2) | 12 (15) | 1 (1) | 1 (1) | 6 (9) | 1 (1) | 1 (1) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Menstruation irregular (Reproductive system and breast disorders) | 0/36 (0) | 0/63 (0) | 0/18 (0) | 0/35 (0) | 0/61 (0) | 1/17 (1) | 0/22 (0) | 0/37 (0) | 0/3 (0) | 0/17 (0) | 0/23 (0) | 0/19 (0) | 0/2 (0) | 0/104 (0) | 0/1 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 0 (0) | 4 (4) | 3 (3) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Maxillofacial operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (3):
  • Study Protocol: RHCD 05 Protocol (b)_Redacted (2018-09-22): https://cdn.clinicaltrials.gov/large-docs/00/NCT03073200/Prot_001.pdf
  • Study Protocol: I1F-MC-RHCD(2.1) Clinical Protocol Addendum (2017-07-20): https://cdn.clinicaltrials.gov/large-docs/00/NCT03073200/Prot_002.pdf
  • Statistical Analysis Plan (2019-06-26): https://cdn.clinicaltrials.gov/large-docs/00/NCT03073200/SAP_000.pdf